CLINICAL TRIAL: NCT03176888
Title: The Efficacy of Reduced-exertion High-intensity Interval Training for Improving Health and Well-being in Newly Diagnosed Female Breast Cancer Patients
Brief Title: Health Benefits of HIT for Breast Cancer Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Logistical problems meant that the study was no longer feasible.
Sponsor: University of Stirling (Other)
Collaborators: University of Bath (Other); Oxford Brookes University (Other)
Responsible Party: Principal Investigator, Niels Vollaard, Principal Investigator, University of Stirling
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2017 0105
Record Dates: First submitted 2017-05-29; First posted 2017-06-06 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Breast Cancer
Keywords: Exercise; Aerobic capacity; Rehabilitation
MeSH Terms: conditions — Breast Neoplasms; Motor Activity | interventions — High-Intensity Interval Training; Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): Patients in the Exercise group will follow a fully-supervised exercise routine (Reduced-exertion, high-intensity interval training (REHIT)) with 3 weekly 10-minute training sessions consisting of easy cycling interspersed with 2 brief 'all-out' cycle sprints. Patients in this group will also be offered up to 6 sessions of cognitive behavioral therapy. The duration of the intervention will be the weeks between enrolling in the study and surgery (~1-4 weeks), as well as an additional period of up to 6 weeks following surgery.
  Interventions: Behavioral: Reduced-exertion, high-intensity interval training (REHIT); Behavioral: Cognitive behavioral therapy (CBT)
- Standard care (No Intervention): Patients allocated to the Standard Care group will receive the care they would have also received if they would not have participated in the study. They will however undergo the same testing sessions as patients in the Exercise group.

INTERVENTIONS:
Behavioral: Reduced-exertion, high-intensity interval training (REHIT) — As in arm/group description
  Arms: Exercise
Behavioral: Cognitive behavioral therapy (CBT) — Up to six 30/40-minute sessions of face-to-face psychotherapy will be offered based on a cognitive model of adjustment to cancer utilizing cognitive and behavioral therapy techniques as described by Moorey & Greer (2012)
  Arms: Exercise

SUMMARY:
Treatment of cancer patients should not only involve removing the cancer, but should also focus on maintaining good health and well-being and quality of life. This can be done by offering patients suitable rehabilitation programmes. Previous research has shown that such programmes need to involve exercise alongside other components, such as psychological support. To date most studies have looked at the positive effects of moderate-intensity exercise such as brisk walking, but this type of exercise is time-consuming and often not done by many patients. Shorter-duration exercise routines consisting of repeated short sprints have been found to improve general health just as well, but one of the most time-efficient routines (termed 'reduced-exertion high-intensity interval training', or 'REHIT') has not been studied in cancer patients. REHIT involves 3 exercise sessions per week, each only 10 minutes long. This makes it an ideal routine to combine with other components of a cancer rehabilitation programme. The present study will determine whether REHIT can improve important markers of health and well-being in newly diagnosed breast cancer patients. To achieve this the investigators will recruit up to 30 patients and divide them into a group who will do REHIT before and for up to 6 weeks after their cancer surgery, and a control group who will receive standard care. Markers of health and well-being will be measured at the start of the study, ~1 week after surgery, and ~7 weeks after surgery. Any changes will be compared between the exercise group and the control group. If beneficial effects are found with the REHIT intervention then this could be more widely implemented as part of cancer treatment. This study is funded by Nuffield Health and will be performed in Oxford, UK.

DETAILED DESCRIPTION:
This study involves a randomised controlled trial: study participants will be randomly allocated to either a group who will receive the care that they would normally have received if they would not have been in the study (control group), and a group who will receive the same standard care but will also be asked to follow a novel supervised exercise routine three times per week before their surgery and for up to 6 weeks after surgery, as well as some psychological support.

Up to 30 newly-diagnosed female breast cancer patients will be recruited. Following written informed consent, participants will be invited for a baseline testing session. This will involve a fasting blood sample (ideally at a time when the patient's medical team would take a blood sample anyway). The investigators will analyse this sample for a number of markers of health, such as blood sugar and fat levels, and markers of inflammation. The investigators will measure the patients' height with a stadiometer, and weight and body fat percentage using a special set of scales. The investigators will ask patients to complete several questionnaires that ask questions about their current well-being. Finally the investigators will measure the patients' handgrip strength as well as their fitness levels. The grip strength test involves squeezing a handheld device as hard as possible for a few seconds. The fitness test involves cycling on a stationary bike with a gradually increasing resistance until the patient cannot continue any longer because of fatigue. In this test the investigators will ask patients to breathe through a tube to determine the maximal amount of oxygen they can take up during exercise. This measure (termed VO2max) is one of the best health markers that can be measured: it is the best predictor of future risk of chronic disease or premature death. All testing sessions will be performed at the Manor Hospital in Oxford (unless the equipment required for the analysis of VO2max is not available for a period of time, in which case patients will be invited to attend Oxford Brookes campus for the fitness test; this is a 4-minute drive from the Manor Hospital).

Ideally, the blood samples will be taken in a fasted state (i.e. in the morning without having had breakfast), whereas the fitness test will be done after the patient has last had some food. The investigators will therefore provide the participants with a light snack after the blood sample has been taken. In case a patient cannot attend the hospital in the morning in a fasted state then they will arrange the session at a later time of day and the patient will not be required to be fasted (leading to loss of some of the secondary outcome measures which require a fasted state).

After the baseline testing has been completed the investigators will tell patients whether they will be in the control group or in the exercise group. Patients in the control group will receive their standard care as if they would not have participated in the study. The research team will not interact with these patients until the second testing session. Patients in the exercise group will be invited to perform 3 fully supervised exercise sessions per week at the Manor Hospital. These exercise sessions will involve 10 minutes of cycling at a low intensity, but with 2 brief cycle sprints after 2 and 6 minutes. The sprints will last 10 seconds in the first week of training, 15 seconds in the second week, and 20 seconds from week 3 onward. Training sessions will be stopped at least 2 days prior to the scheduled surgery date.

Surgery will interrupt the exercise programme. Between 7 and 10 days post-surgery, or when the consultant breast surgeon deems appropriate, all patients will undergo post-surgery testing. Testing procedures will be identical as those for baseline testing.

Following post-surgery testing, patients in the exercise group will resume the exercise programme. The duration of the sprints will restart at 10 seconds in the first week, 15 seconds in the second week, and 20 seconds in the remaining weeks. The exercise routine will be continued until follow-up treatment or for a period of up to 6 weeks. Before or after one of the 3 weekly exercise sessions, patients will receive a 30/40-minute face-to-face session with a psychologist. The aim of these sessions will be to reduce emotional distress, improve mental adjustment, promote a sense of personal control over current experience, develop effective coping strategies for dealing with cancer-related difficulties, and open expression of emotion. If patients cannot attend psychological support sessions then they will be offered the opportunity to catch up through a session over the phone.

Approximately 3 days following the final training session patients will undergo end-of-trial testing, identical to the previous two testing sessions. Patients in the control group will undergo this testing session at a time-point equivalent to that of patients in the exercise group.

ELIGIBILITY:
Inclusion Criteria:

1. Recent diagnosis of biopsy-proven primary invasive breast cancer
2. Pre- or post-menopausal women
3. World Health Organisation Performance status 0-2
4. No distant metastasis
5. On a treatment plan of:

   1. surgery (breast conservation surgery or mastectomy with or without reconstruction, including axillary surgery)
   2. Adjuvant treatment with hormonal therapy and/or radiotherapy
   3. Adjuvant chemotherapy with or without anti-Her-2 therapy
6. Can start the study within 1 week of diagnosis and prior to surgery
7. Have surgery arranged within 1-4 weeks of diagnosis
8. All receptor statuses are eligible

Exclusion Criteria:

1. BMI > 35 kg·m-2
2. Age < 35 y or > 60 y
3. Men
4. Verbal self-report of undertaking five or more structured exercise sessions per week, perceived as being moderate-to-vigorous intensity, and each session being ≥ 30 minutes in duration
5. Contraindications to exercise as determined using the Physical Activity Readiness Questionnaire (PAR-Q)
6. Any known significant cardiovascular (except controlled hypertension), pulmonary (except treated/controlled asthma) or metabolic disease (except hypercholesterolemia or type II diabetes)
7. Auto-immune disease or exercise-limiting inflammatory arthritis
8. Distant metastasis
9. Secondary breast cancer or previous diagnosis of invasive cancer and treatment within last 5 years except

   1. Localised basal cell carcinoma or squamous cell carcinoma of skin
   2. In situ melanoma
   3. Cervical intraepithelial neoplasia (CIN)
10. Neoadjuvant chemotherapy

Ages: 35 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Change in maximal aerobic capacity (VO2max) | From baseline, to 1 week post-surgery and 7 weeks post-surgery.
  VO2max is a measure of the maximal amount of exercise that can be consumed and used during exercise. It is one of the best predictors of future risk of morbidity and mortality. An increase in VO2max represents a positive change in health. The primary outcome measure is change in VO2max from baseline to 1 week post-surgery and 7 weeks post-surgery.

SECONDARY OUTCOMES:
Change in homeostatic model assessment of insulin resistance (HOMA-IR) | From baseline, to 1 week post-surgery and 7 weeks post-surgery.
  HOMA-IR is a measure of risk of type 2 diabetes and metabolic disease.
Change in blood lipid profile | From baseline, to 1 week post-surgery and 7 weeks post-surgery.
  This includes circulating levels of total cholesterol, HDL cholesterol, LDL cholesterol, and triglycerides. These are common health markers.
Change in blood pressure | From baseline, to 1 week post-surgery and 7 weeks post-surgery.
  Blood pressure is a common health marker.
Change in body mass index (BMI) | From baseline, to 1 week post-surgery and 7 weeks post-surgery.
  Height and weight will be measured to calculate BMI (in kg/m^2). BMI is a common health marker.
Change in grip strength | From baseline, to 1 week post-surgery and 7 weeks post-surgery.
  Maximal isometric grip strength assesses how hard a person can squeeze their fist. This is a good marker of risk of future morbidity.
Change in mental well-being | From baseline, to 1 week post-surgery and 7 weeks post-surgery.
  Questionnaires will be used to determine changes in mental well-being.
Change in body fat percentage | From baseline, to 1 week post-surgery and 7 weeks post-surgery.
  Body fat percentage (as determined using bioimpedance scales) is a common health measure.

CONTACTS AND LOCATIONS:
Overall Officials: Niels BJ Vollaard, PhD, Principal Investigator — University of Stirling
Locations (1):
- Manor Hospital, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No
This is a small study which will generate pilot data for larger trials. Although the investigators will publish group data there is no plan to share individual data with other researchers. However, any requests for anonymised individual data will be considered on a case-by-case basis.